CLINICAL TRIAL: NCT06525688
Title: Identification of New Biomarkers and Potential Therapeutic Targets in Clinical Osteoporosis Using Omics Technologies
Brief Title: New Biomarkers and Therapeutic Targets in Osteoporosis Via Omics Technologies
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: National Hellenic Research Foundation (Other)
Responsible Party: Principal Investigator, EFSTATHIOS CHRONOPOULOS, Professor in Orthopedics at National and Kapodistrian University of Athens, Laboratory for Research of the Musculoskeletal System Director, National and Kapodistrian University of Athens
Other Study IDs: 31274/03.07.2024
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis Fracture; Osteoporosis, Severe
Keywords: Osteoporosis; Osteoarthritis; Hip fracture; Postmenopausal Osteoporosis; Proteomics; Metabolomics; Osteoporotic Hip Fracture
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporotic Fractures; Osteoporosis; Osteoarthritis; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bone,Serum and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postmenopausal Female Patient with subcapital hip osteoporotic fracture: Postmenopausal Female Patient with subcapital hip osteoporotic fracture
  Interventions: Other: Bone, Serum and Plasma sample
- Postmenopausal Female Patient with hip osteoarthritis: Postmenopausal female patient with hip osteoarthritis who will undergo total hip replacement.
  Interventions: Other: Bone, Serum and Plasma sample

INTERVENTIONS:
Other: Bone, Serum and Plasma sample — Intervention: Bone samples will be collected during surgery from the femoral neck (which is typically removed and discarded in these operations) and fasting morning blood samples.

SUMMARY:
This study aims to discover novel biomarkers and therapeutic targets for osteoporosis through the use of advanced omics technologies, including proteomics and metabolomics. By analyzing bone and plasma samples from patients with osteoporosis, the research seeks to understand the underlying mechanisms of the disease and identify potential diagnostic and therapeutic biomarkers.

DETAILED DESCRIPTION:
Study Objectives:

1. To investigate the proteomic profile of bone and plasma in clinical osteoporosis compared to patients with osteoarthritis.
2. To study the metabolomic profile of serum in clinical osteoporosis compared to patients with osteoarthriti.
3. To identify and validate potential biomarkers for osteoporosis diagnosis and treatment.
4. To elucidate the pathophysiological mechanisms involved in osteoporosis.

Methodology:

Clinical Osteoporosis:

Patient Recruitment: 60 postmenopausal women will be divided into two groups: those with osteoporotic hip fractures and a control group with osteoarthritis undergoing total hip replacement.

Sample Collection:

Bone Samples: Collected from the femoral neck during surgery, cleaned, and divided into four parts. One part will be used for bone density analysis (pQCT or DXA), and the other parts will be stored for proteomic analysis.

Blood Samples: Fasting morning blood samples will be collected for general biochemical tests, bone turnover markers, and stored for metabolomic and proteomic analyses.

Technologies and Analysis:

Proteomics: Utilizes mass spectrometry to identify and quantify proteins in bone and plasma. Key pathways and protein networks involved in osteoporosis will be identified using bioinformatics tools.

Metabolomics: Analyzes small molecules in serum to uncover metabolic changes associated with osteoporosis. Both targeted and non-targeted approaches will be used to identify significant biomarkers.

Expected Outcomes:

1. Identification of specific proteins and metabolites as biomarkers for osteoporosis.
2. Enhanced understanding of the molecular mechanisms driving bone loss.
3. Validation of therapeutic targets for potential treatment strategies.

Significance:

This integrative approach combining proteomics and metabolomics aims to provide a comprehensive understanding of osteoporosis, facilitating the development of more accurate diagnostic tools and effective treatments for this widespread bone disease.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Female Patients with osteoporotic subcapital femoral neck fracture (Arm 1)
* Postmenopausal Female Patients with hip osteoarthritis that will undergo Total Hip Replacement (Arm 2)

Exclusion Criteria:

* Patients that have undergone before osteoporotic fractures
* Patients with severe cardiovascular, pulmonary, autoimmune, or urinary system conditions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only postmenopausal female patients
Study Population: * Postmenopausal Female Patients with osteoporotic subcapital femoral neck fracture (Arm 1)
  * Postmenopausal Female Patients with hip osteoarthritis that will undergo Total Hip Replacement (Arm 2)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Identification of Proteomic Biomarkers | Up to 18 months.
  The number of proteins identified through proteomic analysis that differ significantly between osteoporosis and control groups
Identification of Metabolomic Biomarkers | Up to 18 months
  The number of small molecules identified through metabolomic analysis that differ significantly between osteoporosis and control groups.

SECONDARY OUTCOMES:
Bone Density Assessment | Up to 18 months
  Bone density measurements using micro-CT in patients with osteoporosis and controls.
Identification of Disrupted Pathways | Up to 18 months
  Analysis of disrupted biological pathways using bioinformatics tools to map the mechanisms affected in osteoporosis.
Correlation of Omics Data with Clinical Markers | Up to 18 months
  Correlation analysis between identified proteomic and metabolomic biomarkers and traditional clinical markers such as CTX and PINP.
Microarchitecture Assessment | Up to 18 months
  Evaluation of bone microarchitecture using histological analysis in osteoporosis patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Chronopoulos, Study Director — KAT General Hospital, Athens Greece
Locations (1):
- Laboratory for Research of the Musculoskeletal System, Kifissia, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
We plan to make individual participant data (IPD) available to other researchers upon reasonable request. Data sharing will be governed by ethical guidelines and privacy regulations to ensure the confidentiality and security of participant information. Interested researchers will be required to submit a formal request, including a brief proposal outlining the intended use of the data. Approved requests will gain access to anonymized data sets, ensuring that participant identities are protected. The aim is to foster collaborative research and maximize the scientific impact of our findings.

DOCUMENTS (1):
  • Study Protocol (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT06525688/Prot_000.pdf